CLINICAL TRIAL: NCT03503591
Title: Post-Market Surveillance Study of the Preceptis Medical, Inc. Hummingbird TTS™ Tympanostomy Tube System
Brief Title: Study of the Hummingbird TTS™ Tympanostomy Tube System
Status: Completed | Type: Observational
Sponsor: Preceptis Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Preceptis PMS
Record Dates: First submitted 2018-04-02; First posted 2018-04-20 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Otitis Media
Keywords: tympanostomy; myringotomy; otitis media; ear tubes; ear infection
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: No

INTERVENTIONS:
Device: Hummingbird Tympanostomy Tube System — Insertion of a ventilation tube under sedation and local anesthetic

SUMMARY:
The objective of this study was continued commercial evaluation of the intraoperative safety and performance of the H-TTS for the placement of ventilation tubes in pediatric patients undergoing a tympanostomy procedure under moderate sedation and local anesthetic.

DETAILED DESCRIPTION:
The study was a multi-site, prospective and retrospective, treatment-only post-market study of the H-TTS. The study was performed in a commercial environment. Patients were already have a scheduled tympanostomy procedure with the H-TTS under moderate sedation and local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months through 5 years of age
* Candidates for ventilation tube placement
* H-TTS used under moderate sedation and local anesthetic

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 6 months through 5 years of age, who are candidates for placement of VT.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Cloud Ear, Nose & Throat, Saint Cloud, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Insertion of a Ventilation Tube Under Sedation and Local Anesthetic: Children 6 months through 5 years of age, who are candidates for placement of VT.
Period: Overall Study
Arm/Group | Insertion of a Ventilation Tube Under Sedation and Local Anesthetic
Started | 109
Completed | 109
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One site enrolled patients prospectively. Data from the other three sites was retrospectively procured from a previous multi-site moderate sedation study using data that was not previously submitted to FDA.
Arm/Group | Insertion of a Ventilation Tube Under Sedation and Local Anesthetic
Number analyzed (Participants) | 109
Age, Continuous [Median (Full Range); unit: Months] | 19 [6 to 57]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex not collected in this study.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Procedures Converted From Sedation to General Anesthesia
Description: Percentage of procedures that require conversion from sedation to general anesthesia
Time Frame: Intra-operative
Measure: Number (95% Confidence Interval); unit: percentage of procedures converted
Arm/Group | Insertion of a Ventilation Tube Under Sedation and Local Anesthetic
Number analyzed (Participants) | 109
percentage of procedures converted | 12.8 [7.9 to 20.6]

2. Primary Outcome: Rate of Intra-operative Adverse Events
Description: Rate of intra-operative adverse events that occur from the beginning to the end of the procedure
Time Frame: Intra-operative
Measure: Number; unit: participants
Arm/Group | Insertion of a Ventilation Tube Under Sedation and Local Anesthetic
Number analyzed (Participants) | 109
participants | 0

3. Primary Outcome: Rate of Adverse Events Through Discharge
Description: Rate of adverse events that occur between the end of the procedure and discharge
Time Frame: Through discharge, estimated to be approximately 90 minutes post-procedure
Measure: Number; unit: percentage of AEs through discharge
Arm/Group | Insertion of a Ventilation Tube Under Sedation and Local Anesthetic
Number analyzed (Participants) | 109
percentage of AEs through discharge | 0

ADVERSE EVENTS:
Time Frame: Intra-operative and pre-discharge
Description: All adverse events (AE) that occured from when the H-TTS entered the ear through discharge were reported. The event type, treatment, severity and relationship of the event to the procedure or to the study device will be assessed by the surgeon.
  Prospective definitions for anticipated adverse events and serious adverse events were included in the protocol attachments. Common occurrences (e.g., minor bleeding, purulent discharge) during a tympanostomy procedure were not considered AEs.
Arm/Group | Insertion of a Ventilation Tube Under Sedation and Local Anesthetic
All-Cause Mortality (participants affected / at risk) | 0/109
Serious Adverse Events (participants affected / at risk) | 0/109
Other Adverse Events (participants affected / at risk) | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03503591/Prot_SAP_000.pdf